CLINICAL TRIAL: NCT00138905
Title: Experimental Study of Mobile Base Station Related Radio-Frequency Electromagnetic Radiation in Healthy Adults and Adolescents
Brief Title: Experimental Study of Mobile Base Station Related Radio-Frequency Electromagnetic Radiation
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Aarhus (Other)
Collaborators: Aalborg University (Other); Aarhus University Hospital (Other)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Prevention
Other Study IDs: 2064-04-0009; Project ID 0402-
Record Dates: First submitted 2005-08-29; First posted 2005-08-30 (Estimated); Last update posted 2007-09-10 (Estimated); Status verified 2007-09

CONDITIONS: Behavior; Cognition Disorders
Keywords: Base station, EMF, human exposure study,Well-being,cognitive
MeSH Terms: conditions — Behavior; Cognition Disorders

INTERVENTIONS:
Device: UMTS mobile basestation radiation

SUMMARY:
The purpose of this study, is to investigate if low intensity electromagnetic radiation, can influence the cognitive performances and well being of healthy adolescents and adults. Furthermore, the purpose is to provide any special information about the subjects which can cause the possible reactions. Finally, the investigation will try to clarify if there is anything specific in the radiation signal that causes the effect

DETAILED DESCRIPTION:
EMF-exposure has been related to reported symptoms of sleep-disorders, headaches, nervousness, fatigue, and concentration difficulties. This study intends to focus on these symptoms related to the UMTS control signal.

The purpose of this study is to investigate the possible annoyance from very low intensity electromagnetic radiation, as it exists from modern antenna masts supporting mobile communication. Also we try to get a better understanding of the specific parts of the signal leading to symptoms. This investigation tries to clarify the risk for both adults and adolescents, other susceptibility factors, and whether the radiation changes cognitive functions. The above mentioned complaints have been related to psychological distress and somatization, and EMF-related complaints have been reported more by individuals with higher somatization tendency. In the present study, we therefore propose to control for symptoms of somatization and personality traits thought to influence perception and reporting of symptoms.

In this study a signal level of 1 volt/meter (2.6 mW/m2) will be used. This level should correspond to the level, experienced by the general public living rather near a base station antenna. The antenna arrangement will produce an approximation to a plane wave, so that the intensity is constant (within 2 dB) over the volume occupied by the subjects. The subjects are required to sit close to a computer screen and keyboard, which will modify the distribution slightly. The climatic chamber used for the study is modified with absorbing lining to dampen reflections from the walls. The chamber is also modified to make it a screened room to prevent external RF fields, and to some extent low frequency fields, to enter the chamber. Except for cables to the keyboard and screen there will be no other electromagnetic radiators in the chamber. The four different exposure types used, are Sham exposure (no radiation from the antennas), a UMTS signal (typical base station signal, 2140 MHz), a CW (continuous wave) of 2140 MHz. and a Wideband W-CDMA signal, f=2140 MHz, modulated with a random data sequence at a chip rate of 3.8 MHz, corresponding to a pure UMTS modulation signal, without the control signals.

ELIGIBILITY:
Inclusion Criteria:

* Healthy Subjects
* Age 15-16 or 25-40 years

Exclusion Criteria:

* Pregnant
* Subjects with current or previous cardiovascular disease
* Subjects with current or previous fractured scull
* Subjects with chronic lung disease
* Subjects with diseases, which could involve a risk for the subject or possibly influence the outcome measurements

Ages: 15 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 80
Dates: Start 2005-02; Study Completion 2006-04 (Actual)

PRIMARY OUTCOMES:
Trail Making B (time in seconds)

SECONDARY OUTCOMES:
Reaction Time (RTI), complex reaction and movement time: time (in seconds);
Rapid Visual Information Processing (RVP), RVP A': score (between 0 and 1);
Paired Associated Learning (PAL), PAL Stages completed: (0, 1, 2, 3, 4, 5, 6)

CONTACTS AND LOCATIONS:
Overall Officials: Jørgen B. Andersen, Prof., Study Director — Aalborg University
Locations (1):
- Dept. of Environmental and Occupational Medicine, Institute of Public Health, University of Aarhus, Vennelyst Boulevard 6. Build. 260., Aarhus C, Denmark